CLINICAL TRIAL: NCT03167346
Title: The Investigation of Public Awareness of Core Stroke Symptoms
Acronym: IPACSS
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bin Peng, Professor, Peking Union Medical College Hospital
Other Study IDs: PUMCH-IPACSS2017
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Awareness; Health Knowledge, Attitudes, Practice; Core Symptoms; FAST
Keywords: stroke; core symptoms; public awareness; FAST
MeSH Terms: conditions — Stroke; Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate public awareness of core stroke symptoms in more than 40 years old population and its related factors.

ELIGIBILITY:
Inclusion Criteria:

* More than 40 years old (born before December 31st 1976) without specific requirements.
* Be able to finish the questionnaire.

Exclusion Criteria:

* Participants with disturbance of consciousness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are more than 40 years old without specific requirements. This study is a population-based screening programme.
Sampling Method: Probability Sample
Enrollment: 243279 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
awareness rate | 2017-2017
  The awareness rate of core symptoms (FAST: facial droop, arm weakness, speech disturbance, time to call an ambulance)

SECONDARY OUTCOMES:
Associated factors | 2017-2017
  The associated factors with the stroke recognition/ correct action to stroke
Subgroup analysis | 2017-2020
  Analysis of stroke recognition rate and correct action rate and their associated factor in subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Peng, Principal Investigator — Department of Neurology,Peking Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Neurology,Peking Union Medical College Hospital,Shuaifuyuan 1,Dong Cheng District. Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wolters FJ, Paul NL, Li L, Rothwell PM; Oxford Vascular Study. Sustained impact of UK FAST-test public education on response to stroke: a population-based time-series study. Int J Stroke. 2015 Oct;10(7):1108-14. doi: 10.1111/ijs.12484. Epub 2015 Apr 8. PMID 25854424
- [Background] Dombrowski SU, White M, Mackintosh JE, Gellert P, Araujo-Soares V, Thomson RG, Rodgers H, Ford GA, Sniehotta FF. The stroke 'Act FAST' campaign: remembered but not understood? Int J Stroke. 2015 Apr;10(3):324-30. doi: 10.1111/ijs.12353. Epub 2014 Aug 6. PMID 25130981
- [Background] Amano T, Yokota C, Sakamoto Y, Shigehatake Y, Inoue Y, Ishigami A, Hagihara T, Tomii Y, Miyashita F, Toyoda K, Minematsu K. Stroke education program of act FAST for junior high school students and their parents. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):1040-5. doi: 10.1016/j.jstrokecerebrovasdis.2013.08.021. Epub 2013 Oct 2. PMID 24094446
- [Background] Jin H, Zhu S, Wei JW, Wang J, Liu M, Wu Y, Wong LK, Cheng Y, Xu E, Yang Q, Anderson CS, Huang Y; ChinaQUEST (Quality Evaluation of Stroke Care and Treatment) Investigators. Factors associated with prehospital delays in the presentation of acute stroke in urban China. Stroke. 2012 Feb;43(2):362-70. doi: 10.1161/STROKEAHA.111.623512. Epub 2012 Jan 12. PMID 22246693
- [Background] Zhao J, Liu R. Stroke 1-2-0: a rapid response programme for stroke in China. Lancet Neurol. 2017 Jan;16(1):27-28. doi: 10.1016/S1474-4422(16)30283-6. Epub 2016 Oct 28. No abstract available. PMID 28029517
- [Background] Longde W, Ling Y, Yang H, Yi Z, Yongjun W, Xunming J, Xiaoyuan N, Qiumin Q, Li H, Yuming X, Mei L, Jiayi S, Jing L, Dong Z. Fixed-dose combination treatment after stroke for secondary prevention in China: a national community-based study. Stroke. 2015 May;46(5):1295-300. doi: 10.1161/STROKEAHA.114.007384. Epub 2015 Mar 17. PMID 25782466
- [Background] Teuschl Y, Brainin M. Stroke education: discrepancies among factors influencing prehospital delay and stroke knowledge. Int J Stroke. 2010 Jun;5(3):187-208. doi: 10.1111/j.1747-4949.2010.00428.x. PMID 20536616
- [Background] Bouckaert M, Lemmens R, Thijs V. Reducing prehospital delay in acute stroke. Nat Rev Neurol. 2009 Sep;5(9):477-83. doi: 10.1038/nrneurol.2009.116. Epub 2009 Aug 11. PMID 19668246
- [Background] Fassbender K, Balucani C, Walter S, Levine SR, Haass A, Grotta J. Streamlining of prehospital stroke management: the golden hour. Lancet Neurol. 2013 Jun;12(6):585-96. doi: 10.1016/S1474-4422(13)70100-5. PMID 23684084